CLINICAL TRIAL: NCT05864963
Title: Medial Tab-type Fasciocutaneous Flap as an Alternative for the Management of Soft Tissue Defects of the Leg
Brief Title: Medial Tab Flap for Soft Tissue Defects of the Leg
Status: Completed | Type: Observational
Sponsor: Fundación Campbell (Other)
Responsible Party: Sponsor
Other Study IDs: FC05052023
Record Dates: First submitted 2023-05-08; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Leg Coverage Defects
Keywords: Lower extremity reconstruction; leg coverage defects; fasciocutaneous flaps; muscular flaps; orthoplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: 18 patients treated with medial tab-type fasciocutaneous flaps
  Interventions: Procedure: Medial tab-type fasciocutaneous flap
- Control group: 46 patients were randomly chosen, through Propensity Score Matching (PSM) the matching was performed with the age variable. The types of flaps considered were: 15 cases with sural flap, 18 with soleus flap, and 13 with a gastrocnemius flap

INTERVENTIONS:
Procedure: Medial tab-type fasciocutaneous flap — The flap can be taken in different ways depending on the defect. Once the base of the flap is identified, the posterior edge of the tibia is taken as reference; marking of the tab is performed considering that the posterior incision is located 5 cm from the posterior edge of the tibia, and the anterior incision is located longitudinally of the medial region of the tibial diaphysis, the length of the incision depends on the base of the flap and the defect's size.
  The posterior incision is made first in the skin, subcutaneous cellular tissue until the fascia is identified; the subfascial flap is dissected to avoid injuring perforators, dissection is completed up to the anterior edge of the flap, if needed direct cutaneous perforators are ligated; once the subfascial plane has been identified and dissected, the tab is completed in its proximal or distal part according to the previous surgical planning. Later, the tab is rotated to the anterior region of the tibia to cover the defect.
  Groups: Intervention group

SUMMARY:
Selecting the right technique for lower limb soft tissue reconstruction is a therapeutic challenge. Despite having several reconstruction options, it's important to choose a technique that is effective and with the least possible donor site morbidity for the patient.

Objective: demonstrate the therapeutic efficacy of the medial tab flap in soft tissue reconstruction on the leg, compared to conventional flaps.

Materials and methods: Cohort study matched with Propensity Score Matching (PSM) by age. 64 patients with soft tissue defects were selected and followed up to one year postoperatively. Outcome variables: surgical time in minutes, healing, healing time in days, complications.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of soft tissue defects in the leg due to grade III B open fractures, or due to bone infection
* contraindication to using conventional flaps due to the following reasons: soft tissue injuries at the flap island site, injury to the vascular bed of the flap or injury of the flap structure (fascia, skin or muscle)
* people between 18 and 70 years of age

Exclusion Criteria:

* Patients with a history of free flaps
* Whose clinical follow up couldn't be completed to assess outcomes were excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 216 patients with soft tissue defects on the anterior aspect of the leg underwent surgery during the study period, of these 18 patients were treated with medial tab-type fasciocutaneous flaps, this group constituted the intervention group. 198 underwent surgery with conventional flaps, of which 46 patients were randomly chosen, through Propensity Score Matching (PSM) the matching was performed with the age variable. The types of flaps considered were: 15 cases with sural flap, 18 with soleus flap, and 13 with a gastrocnemius flap
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Differences in surgical and healing time between medial tab flaps and conventional flaps | January 2019 - December 2022
  This information was taken from he Sculapio software clinical records, the surgical time was measured in minutes from the moment of the incision to the clousure of the surgical planes, and the healing time was measured in days from the immediate postoperative period until the wound epithelization

SECONDARY OUTCOMES:
Sociodemographic and clinical characteristics | January 2019 - December 2022
  The data collection was made from the Sculapio software clinical records of the Fundacion Campbell
Complications | January 2019 - December 2022
  The complications were descripted from the clinic history recorded by the orthopedic surgeon specialist, the following pathologies were taken into account: necrosis, suture dehiscence, fistula, foreign body granuloma, enlargement of the defect and infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacion Campbell, Barranquilla, Atlántico, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh A, Jiong Hao JT, Wei DT, Liang CW, Murphy D, Thambiah J, Han CY. Gustilo IIIB Open Tibial Fractures: An Analysis of Infection and Nonunion Rates. Indian J Orthop. 2018 Jul-Aug;52(4):406-410. doi: 10.4103/ortho.IJOrtho_369_16. PMID 30078900
- [Background] Parrett Brian M, Pribaz Julian J. Reconstrucción de extremidad inferior. Rev Médica Clínica Las Condes. 2010;21(1):76-85
- [Background] Rodríguez Lara JN, Ochoa Fletes MP. Serie de casos: colgajo sóleo-gastrocnemio en pacientes con defectos de partes blandas en miembros inferiores. Rev Med Hondur. 2021;89(2):131-6
- [Background] Martinov M, Argirova M. Fasciocutaneous flaps in the lower limb soft tissue reconstruction - A surgical case series. Orthoplastic Surg [Internet]. 2022;9(May):1-8. Available from: https://doi.org/10.1016/j.orthop.2022.05.002
- [Background] Friedrich JB, Katolik LI, Hanel DP. Reconstruction of soft-tissue injury associated with lower extremity fracture. J Am Acad Orthop Surg. 2011 Feb;19(2):81-90. doi: 10.5435/00124635-201102000-00003. PMID 21292931
- [Background] Vergara-amador E. El uso de colgajos en la reconstrucción de defectos de cobertura en la pierna distal y dorso de pie The use of flaps in the reconstruction of defects of coverage in the distal leg and dorsum of the foots. 2013;29(1):74-82.
- [Background] MacKechnie MC, Flores MJ, Giordano V, Terry MJ, Garuz M, Lee N, Padilla Rojas LG, MacKechnie MA, Bidolegui F, Brown K, Quintero JE, Ding A, Sanchez Valenciano CG, Tabares Neyra H, Segovia J, Aguilar D, van Lieshout EM, Verhofstad MH, Miclau T. Management of soft-tissue coverage of open tibia fractures in Latin America: Techniques, timing, and resources. Injury. 2022 Apr;53(4):1422-1429. doi: 10.1016/j.injury.2022.01.027. Epub 2022 Jan 19. PMID 35101259
- [Background] Taylor GI, Palmer JH. The vascular territories (angiosomes) of the body: experimental study and clinical applications. Br J Plast Surg. 1987 Mar;40(2):113-41. doi: 10.1016/0007-1226(87)90185-8. PMID 3567445
- [Background] Attinger CE, Evans KK, Bulan E, Blume P, Cooper P. Angiosomes of the foot and ankle and clinical implications for limb salvage: reconstruction, incisions, and revascularization. Plast Reconstr Surg. 2006 Jun;117(7 Suppl):261S-293S. doi: 10.1097/01.prs.0000222582.84385.54. PMID 16799395
- [Background] Concha JM, Camaro PL, David A, Concha C. The lateral supramalleolar flap for the treatment of open foot and ankle fractures. Orthoplastic Surg [Internet]. 2022;9(May):80-5. Available from: https://doi.org/10.1016/j.orthop.2022.07.006
- [Background] Mahajan RK, Srinivasan K, Singh M, Jain A, Kapadia T, Tambotra A. Management of Post-Traumatic Composite Bone and Soft Tissue Defect of Leg. Indian J Plast Surg. 2019 Jan;52(1):45-54. doi: 10.1055/s-0039-1688097. Epub 2019 May 8. PMID 31456612
- [Background] Luo Z, Dong Z, Ni J, Wei J, Peng P, Lv G. Distally Based Peroneal Artery Perforator-Plus Fasciocutaneous Flap to Reconstruct Soft Tissue Defect Combined With Chronic Osteomyelitis in the Lateral Malleolus. Int J Low Extrem Wounds. 2022 Dec;21(4):464-470. doi: 10.1177/1534734620956782. Epub 2020 Sep 11. PMID 32912022
- [Background] Akhtar S, Hameed A. Versatility of the sural fasciocutaneous flap in the coverage of lower third leg and hind foot defects. J Plast Reconstr Aesthet Surg. 2006;59(8):839-45. doi: 10.1016/j.bjps.2005.12.009. Epub 2006 Mar 9. PMID 16876082
- [Background] Economides JM, DeFazio MV, Golshani K, Cinque M, Anghel EL, Attinger CE, Evans KK. Systematic Review and Comparative Meta-Analysis of Outcomes Following Pedicled Muscle versus Fasciocutaneous Flap Coverage for Complex Periprosthetic Wounds in Patients with Total Knee Arthroplasty. Arch Plast Surg. 2017 Mar;44(2):124-135. doi: 10.5999/aps.2017.44.2.124. Epub 2017 Mar 15. PMID 28352601
- [Background] Zweifel-Schlatter M, Haug M, Schaefer DJ, Wolfinger E, Ochsner P, Pierer G. Free fasciocutaneous flaps in the treatment of chronic osteomyelitis of the tibia: a retrospective study. J Reconstr Microsurg. 2006 Jan;22(1):41-7. doi: 10.1055/s-2006-931906. PMID 16425121
- [Background] Roberts HJ, DeSilva GL. Can Sural Fasciocutaneous Flaps Be Effective in Patients Older Than 65? Clin Orthop Relat Res. 2020 Apr;478(4):734-738. doi: 10.1097/CORR.0000000000000963. PMID 32229743
- [Background] Dhamangaonkar AC, Patankar HS. Reverse sural fasciocutaneous flap with a cutaneous pedicle to cover distal lower limb soft tissue defects: experience of 109 clinical cases. J Orthop Traumatol. 2014 Sep;15(3):225-9. doi: 10.1007/s10195-014-0304-0. Epub 2014 Jun 24. PMID 24957508
- [Background] Donski PK, Fogdestam I. Distally based fasciocutaneous flap from the sural region. A preliminary report. Scand J Plast Reconstr Surg. 1983;17(3):191-6. doi: 10.3109/02844318309013118. PMID 6673085
- [Background] Wee JT. Reconstruction of the lower leg and foot with the reverse-pedicled anterior tibial flap: preliminary report of a new fasciocutaneous flap. Br J Plast Surg. 1986 Jul;39(3):327-37. doi: 10.1016/0007-1226(86)90042-1. PMID 3730678
- [Background] Erdmann MW, Court-Brown CM, Quaba AA. A five year review of islanded distally based fasciocutaneous flaps on the lower limb. Br J Plast Surg. 1997 Sep;50(6):421-7. doi: 10.1016/s0007-1226(97)90329-5. PMID 9326145
- [Background] Bullocks JM, Hickey RM, Basu CB, Hollier LH, Kim JY. Single-stage reconstruction of Achilles tendon injuries and distal lower extremity soft tissue defects with the reverse sural fasciocutaneous flap. J Plast Reconstr Aesthet Surg. 2008;61(5):566-72. doi: 10.1016/j.bjps.2006.01.017. Epub 2007 Mar 26. PMID 17369010